CLINICAL TRIAL: NCT06284252
Title: The Effect of Virtual Game Simulation on Nursing Students' Physical Examination Skills for the Heart, Abdomen and Respiratory System: Randomized Controlled Study
Brief Title: Virtual Game Simulation on Nursing Students' Physical Examination Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: TÜBİTAK-323S135
Record Dates: First submitted 2024-02-15; First posted 2024-02-28 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Simulation of Physical Illness
Keywords: Virtual Gamin Simulation; Nursing Students; Physical Examination

STUDY DESIGN:
Intervention Model Description: Control group and intervention group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant blinding: In order to ensure participant blinding, all students will register to the site where virtual game simulations will be hosted.
  Statistics blinding: In order to blind the statistics expert, at the end of data collection, the website expert will share the collected data with the statistics expert as group A and B data. The statistician will perform statistical analyzes without knowing which group is the control and which group is the experiment.
  Researcher blinding: In order to ensure researcher blinding, the expert who designed the web page for virtual game simulations selected the students who registered on the website, using the "A" and "B" codes, according to the list he received from the statistics expert, on the website with a random group as control and one group as experiment. will assign it to the site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This is the group that takes theoretical lessons and does not play virtual games. Students will receive physical examination training and participate in laboratory practices. Pre-test and post-test skill evaluation will be made.
- Initiative group (Experimental): Students will participate in theoretical training and laboratory practice. Students will play three different virtual game simulations. Students will participate in pre-test and post-test skill practice.
  Interventions: Other: Virtual Gaming Simulation

INTERVENTIONS:
Other: Virtual Gaming Simulation — Two-dimensional virtual game simulations that can be played on computers will be developed using the recorded videos. Games will focus on physical examination of the heart, abdomen and respiratory system. The developed games will be played to the intervention group.
  Arms: Initiative group

SUMMARY:
The project is unique in that it will use virtual game simulation, a new learning method, and it will address the physical examination skills of nursing students, an area that has not been researched before. In the project, a randomized controlled research design with a pretest-posttest control group will be used. The population will consist of 200 second-year students enrolled in the Physical Examination in Nursing course at Necmettin Erbakan University, Faculty of Nursing, Department of Nursing, in the 2024-2025 Fall Semester. 120 students from the population who meet the research inclusion criteria will be randomly assigned to control (n=60) and experimental (n=60) groups according to their general academic success score. In collecting data; Introductory characteristics form, skill checklist for physical examination of the heart, skill checklist for physical examination of the abdomen, skill checklist for physical examination of the respiratory system and an evaluation form for the effect of virtual game simulation on skill practice for physical examination will be used. In the project, three different virtual game simulations will be developed for physical examinations of the heart, abdomen and respiratory system. During the fall semester, theoretical and laboratory demonstration applications will be carried out by the project team. A pre-test will be administered to all students, and then virtual game simulations will be made available to students in the experimental group for three weeks. Then, the virtual games will be closed to the students and a post-test will be administered to the experimental and control group students. After the final test application, virtual game simulations will be made available to students in the control group. In pre- and post-test applications, students will practice physical examination skills on simulated patients at three different stations (heart, abdomen and respiratory system) and will be evaluated by the project team according to skill checklists. After the skill evaluations, the students in the experimental group will be given a form to evaluate the effect of the virtual game simulation for physical examination on skill practice and will be asked to fill it out.

DETAILED DESCRIPTION:
One of the most important components in providing professional and holistic nursing care is health assessment. Assessment of the individual's health status consists of three stages: history taking, physical examination and recording of data. The first step in providing safe and effective nursing care is to use physical examination skills. Physical examination is a systematic data collection method obtained by using the methods of inspection (visual examination), palpation (hand examination), auscultation (examination by listening), percussion (examination by hitting) and olfaction (examination by smell) in order to determine the health problems of the individual.

Physical examination helps determine changes in the patient's health status, provide systematic holistic nursing care, plan care with data obtained as a result of comprehensive and objective measurements, and make effective decisions regarding the individual's health status. Depending on the developments in nursing roles, nurses are now responsible for performing physical examinations.

In clinical practice, physical examination skills are used to measure an individual's vital signs, determine height and body weight, and evaluate skin integrity, extremity movements, and bowel movements in the early postoperative period. However, in order to make a comprehensive evaluation and collect objective data, physical examination skills should be used more effectively and this issue should be emphasized in nursing education. West (2006) states that physical examination should be included in nursing education to establish a connection between symptoms and physiology, contribute to the quality of care, and ensure strong collaboration with other health professionals. However, research shows that physical examination methods are not emphasized enough in undergraduate nursing courses. In addition, it was determined that nurses and students did not widely use physical assessment methods in practice. These examination methods are not adequately offered to nursing students because physical evaluation is included in the elective course that many universities do not offer. Doğdu et al. (2021) barriers to nursing students using physical examination methods; They stated this as corporate culture, lack of time, knowledge and skills. Therefore, it is necessary to provide students with physical examination knowledge and skills in nursing education.

It is stated in the literature that the skill that students have the most difficulty in learning is respiratory system examination, especially auscultation skill. In a study, 177 educators were asked about the physical examination skills that should be taught first and they stated that the level of consciousness, heart, abdomen and respiratory system examination should be taught first. In another study, students stated that they frequently performed heart, abdomen and lung examinations in clinical practice, but most of the students stated that they did not perform a complete physical examination and that the practice was not sufficient.This project aims to teach physical examination skills for the heart, abdomen and respiratory system, which students frequently encounter in clinical practice and have difficulty in practicing skills.

It is very difficult to teach physical examination skills to students with classical learning methods. Today, with the propensity of Generation Z students towards information technologies, classical learning methods and teaching methods that include technology have begun to be used together.

Recently, one of the teaching methods that incorporate technology in nursing education is virtual game simulation. Virtual game simulation is a two-dimensional (2D) virtual computer game involving simulated people that enables students to actively participate in a clinical scenario. Virtual game simulations are a pedagogical method that allows students to use critical thinking and decision-making skills by using simulated patients in scenarios involving different clinical environments.

Studies have been conducted with nursing students using virtual game simulations in the fields of obstetrics, pediatrics, geriatrics, mental health, surgery, respiratory system diseases, emergency health and nursing process, and in these studies, virtual game simulation has been shown to improve students' knowledge, feedback, interaction, participation, self-confidence, self-efficacy. It is stated that it increases perception, satisfaction, critical thinking, decision-making skills, learning and psychomotor skills. In studies, nursing students stated that virtual game simulations are usable, easy, fun and useful, reduce clinical anxiety, increase their self-confidence, self-efficacy and memorability, and allow learning and practice in a safe, realistic and interesting environment. It is also stated that virtual game simulation is very useful for nursing students (Atthill et al. 2021; Luctkar-Flude et al. 2021; Verkuyl et al. 2021). However, since virtual game simulation is a new learning method, there is only one experimental study examining its effect on the skill level of nursing students. In this study, it was determined that virtual game simulation increased the general performance scores of nursing students (n = 20) regarding resuscitation. Virtual game simulation can be used in teaching physical examination skills, which is one of the professional practices of nursing.

ELIGIBILITY:
Inclusion Criteria:

* Taking the Physical Examination course in Nursing for the first time,
* Having access to the Internet,
* Volunteering to participate in the research.

Exclusion Criteria:

* Not participating in in-class and out-of-class processes regarding the heart, abdomen and respiratory system,
* Not participating in one of the steps of the research (pre-test, playing virtual game simulations, post-test)
* Wants to leave the research.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Skill assessment for physical examination of the abdomen (Pretest) | up to 9 months
  Skills Checklist for Physical Examination of the Abdomen
Skill assessment for physical examination of the heart(Pretest) | up to 9 months
  Skills Checklist for Physical Examination of the Heart
Evaluation of physical examination skills of the respiratory system(Pretest) | up to 9 months
  Skills Checklist for Physical Examination of the Respiratory System

SECONDARY OUTCOMES:
Skill assessment for physical examination of the abdomen (Posttest) | up to 11 months
  Skills Checklist for Physical Examination of the Abdomen
Skill assessment for physical examination of the heart(Posttest) | up to 11 months
  Skills Checklist for Physical Examination of the Heart
Evaluation of physical examination skills of the respiratory system(Posttest) | up to 11 months
  Skills Checklist for Physical Examination of the Respiratory System

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)